CLINICAL TRIAL: NCT06354101
Title: The VITALITY Registry
Brief Title: The Purpose of This Registry Study is to Learn More About Metabolic Health: Approximately 15,000 Participants Who Are Overweight or Have Obesity With or Without Metabolic Diseases Are Expected to Participate in This Registry Study.
Status: Withdrawn | Type: Observational
Why Stopped: Terminated by sponsor before enrolling any patients into the study.
Sponsor: CorEvitas (Network)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CorEvitas-VITALITY
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-03

CONDITIONS: Metabolic Health
MeSH Terms: interventions — Tirzepatide; semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Tirzepatide — Once-weekly subcutaneous injectable
Drug: Semaglutide — Once-weekly subcutaneous injectable

SUMMARY:
The purpose of this registry study is to learn more about metabolic health. The information gathered will be used to support research on the natural history of obesity and weight related diseases, their treatments, and how it affects overall health. Approximately 15,000 participants who are overweight or have obesity with or without metabolic diseases are expected to participate in this registry study.

DETAILED DESCRIPTION:
The VITALITY Registry is a research study to collect healthcare information on people with conditions related to their weight which is stored in a database. Participants, along with their doctor, provide the health information that makes up this database. Participants will not be asked to take any special treatments or tests as part of the study.

Participants will be asked to complete questionnaires 2 times a year for up to 10 years, and the doctor will be asked to enter certain available information from office visits 1 time per year for up to 10 years regarding health, treatments, and symptoms related to the participants metabolic health.

The information that will be collected for this study will include demographics (for example, age, gender, race, employment, etc.), medical history (including all prior and current treatments), social history, details about your metabolic health, how metabolic health impacts daily life, mental health, and satisfaction with treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age (or age of majority)
* Willing to provide consent to participate

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, observational registry to study metabolic health in individuals.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Main Objective of Registry | Up to 10 years
  The main objective of the registry is real-world evidence reflecting the experience of individuals in regards to their metabolic health.

IPD SHARING:
Plan to Share IPD: No